CLINICAL TRIAL: NCT02500875
Title: Treatment of Infected Surgical Wounds With Negative Pressure Topical Therapy and Instillation (With or Without Antiseptic) Versus no Instillation
Acronym: PTN-INSTILL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associazione Infermieristica per lo studio delle Lesioni Cutanee (Other)
Responsible Party: Principal Investigator, Gabrielli Barbara, Physician, Associazione Infermieristica per lo studio delle Lesioni Cutanee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AISLeC-004
Record Dates: First submitted 2015-05-24; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-05

CONDITIONS: Infected Surgical Wound
Keywords: Negative-Pressure Wound Therapy; Topical Negative Pressure Therapy; Sodium Hypochlorite
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PTNiA (Experimental): Topical negative pressure therapy with instillation of saline solution (6 times daily).
  During the instillation of saline solution, aspiration is stopped for 10-15 minutes and subsequently the device is programmed to exert a sub atmospheric pressure in aspiration of at least 50 mmHg up to a maximum of 200 mmHg.
  The change of dressing is carried out on the first day after the application of the device, and thereafter, as needed (approximately every 3 or 4 days).
  Interventions: Device: PTNiA
- PTNiB (Experimental): Topical negative pressure therapy with instillation of Amukine Med 0,05% (6 times daily).
  During the instillation of Amukine Med 0,05%, aspiration is stopped for 10-15 minutes and subsequently the device is programmed to exert a sub atmospheric pressure in aspiration of at least 50 mmHg up to a maximum of 200 mmHg.
  The change of dressing is carried out on the first day after the application of the device, and thereafter, as needed (approximately every 3 or 4 days).
  Interventions: Device: PTNiB
- PTN (Active Comparator): Topical negative pressure therapy (without instillation). The device is programmed to exert a sub atmospheric pressure in aspiration of at least 50 mmHg up to a maximum of 200 mmHg.
  The change of dressing is carried out on the first day after the application of the device, and thereafter, as needed (approximately every 3 or 4 days).
  Interventions: Device: PTN

INTERVENTIONS:
Device: PTNiA
  Arms: PTNiA
Device: PTNiB
  Arms: PTNiB
Device: PTN
  Arms: PTN

SUMMARY:
The objective of this study is to evaluate the effectiveness of PTNi therapy versus PTN therapy without instillation in the treatment of infected surgical wounds. Investigators mean to verify differences of effectiveness between the different types of instilled substances, normal saline versus Amukine Med 0.5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with infected surgical wounds.
* Patient age greater than or equal to 18 years.
* Patients who have given informed consent to the enrollment in the trial and to the processing of personal data.

Exclusion Criteria:

* Patients unable of consent.
* Patients affected by serious medical conditions that, according to the investigator's opinion, represent a contraindication to the study participation.
* Patients affected by wounds with exposition of blood vessels, sutures, organs or nerves and open wounds in mediastinum or abdomen.
* Patients with malignancy at the wound.
* Patients with untreated osteomyelitis.
* Patients with enteric and unexplored fistulas.
* Patients with necrotic tissue and eschar.
* Immunocompromised patients or in treatment with corticosteroids.
* Suspected or known allergic diathesis to the product of medication.
* Patients with coagulation disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Absence of clinical infection (according NHSN 2014) | 1 month
  frequency of wound without clinical infection
Absence of clinical infection | 1 month
  number of days to absence clinical infection

SECONDARY OUTCOMES:
Treatment days | 1 month
  number of days to wounds treatment
Wound closure | 1 month
  number of days to wounds closure
Patient's discharge | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  number of days to patient's discharge
Patient's pain (Numeric Rating Scale (NRS) | 1 month
  assessment with Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Chiari, Principal Investigator — Policlinico Sant'Orsola Malpighi Bologna
Locations (1):
- Policlinico Sant'Orsola Malpighi, Bologna, Bologna, Italy